CLINICAL TRIAL: NCT05636280
Title: Evaluation of the Effect of Three Dimensional Schroth Exercises on Abdominal Muscle Thickness in Patients With Adolescent Idiopathic Scoliosis
Brief Title: The Effect of Schroth Exercises on Abdominal Muscle Thickness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Zeynep Ayyıldız Eroğlu, MSc Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Schroth Intervention
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Scoliosis Idiopathic
Keywords: scoliosis; abdominal muscle thickness; schroth exercise
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- schroth exercise group (Experimental): In this study, Schroth exercise training applied 3 days a week for 6 weeks in people with Adolescent Idiopathic Scoliosis will be applied by a physiotherapist trained in schroth.
  Interventions: Other: schroth exercise
- traditional scoliosis exercise group (Active Comparator): In this study, traditional scoliosis exercise training applied 3 days a week for 6 weeks in people with Adolescent Idiopathic Scoliosis will be applied by a physiotherapist.
  Interventions: Other: traditional scoliosis exercise

INTERVENTIONS:
Other: schroth exercise — In this study, Schroth exercise training applied 3 days a week for 6 weeks in people with Adolescent Idiopathic Scoliosis will be applied by a physiotherapist trained in schroth.
  Arms: schroth exercise group
Other: traditional scoliosis exercise — In this study, traditional scoliosis exercise training applied 3 days a week for 6 weeks in people with Adolescent Idiopathic Scoliosis will be applied by a physiotherapist.
  Arms: traditional scoliosis exercise group

SUMMARY:
Although abdominal muscle thickness has been evaluated in individuals with scoliosis in the literature, there is no study in the literature reporting the relationship between abdominal muscle thickness under ultrasound as a result of schroth exercises. The aim of this study is to evaluate the effectiveness of the Schroth method on abdominal muscle thickness in people with AIS.

DETAILED DESCRIPTION:
Scoliosis is defined as the lateral curvature of the spine more than 10 degrees to the right or left, detected radiologically in the coronal plane, but scoliosis is a complex three-dimensional orthopedic deformity that also affects the spine, shoulder girdle and pelvis. The etiopathogenesis of scoliosis is still unclear and the cause cannot be determined in 80% of cases, and it is called idiopathic scoliosis. Other causes include neurological, bone origin, trauma, joint and connective tissue pathologies. Scoliosis causes postural changes in the whole body of the person due to the rotation and angulation of the spine. Especially the abdominal muscles, rib cage, back and waist extensors are most affected by this condition, and it causes biomechanical changes in the pelvis, shoulder girdle and even lower extremities and feet. The spine causes severe morphological changes due to vertebral wedging and rib cage distortion. Vertebral wedging causes a progressive vertebral deformation associated with axial rotation and scoliosis progression. This vertebral deformation is not only associated with the deterioration of the bone structure and the spine, but also causes changes in the structures of the upper extremity and lower extremity. In the treatment of scoliosis; There are four main categories as observation, corset, physiotherapy and rehabilitation applications and surgery. These treatments should be decided by considering the risk of curvature progression. The main purpose in the treatment of scoliosis is to prevent curvature progression. In scoliosis, besides the spine, shoulder girdle, trunk muscles, pelvis and even lower extremities are also affected by this pathological condition and postural problems occur. Therefore, a detailed clinical analysis and evaluation of the entire musculoskeletal system should be performed in individuals with scoliosis. The problem is determined by revealing in detail the length, strength and functional status of the muscles and ligaments that cause impaired body cosmetics. It has been reported in the literature that pelvic anomalies occur with the progression of scoliosis. Qui et al. reported that there is a difference between the right and left of the pelvis, which is not due to developmental asymmetry or distortion of the pelvis, but due to horizontal rotation. At the same time, Gum et al. reported that people with adolescent idiopathic scoliosis (AIS) have advanced pelvic rotations in the transverse plane. Panjabi et al. reported that the system model of the spine consists of passive, active and control subsystems. Any problem that may occur in these three systems is compensated by other systems responsible for carrying out coordinated activities. trunk muscles; especially the multifidus, transverse abdominus and internal obliques are examples of active systems. Contraction of these muscles plays an important role in trunk stabilization by increasing abdominal pressure and elongation of the thoracolumbar fascia. In the magnetic resonance imaging study conducted with people with AIS, changes were observed in the type 2 fibers of the multifidus muscle on the concave side of the apex of the curve. The European Society of Scoliosis Orthopedics and Rehabilitation (SOSORT) recommends scoliosis-specific exercises in addition to bracing for scoliosis. It has been reported that the progression of the curve is very rapid if there is a progression of 5.4 degrees and above in the measurements taken every 6 months for curves of 25 degrees and above and these people should be included in the treatment. Although bracing is a difficult treatment to accept in some children, the acceptance of exercise therapy is higher. Schroth exercises are specialized exercises for scoliosis and have been reported to reduce the Cobb angle of curvature, improve neuromotor control, increase respiratory function and back flexibility, and improve cosmetic appearance. The Schroth method includes scoliosis-specific sensorimotor, posture and breathing exercises, and provides the prevention of 3-dimensional spinal deformities in the spine by the formation of postural realignment in people with AIS. With the autocorrection included in the method, self-elongation and postural correction are provided to each curvature pattern and the person's muscle imbalance is balanced. It has been reported that with Schroth exercises, muscle strength and flexibility are increased, the Cobb angle is improved, and surgery rates are reduced. Kim et al., in their study in which they examined the abdominal muscle thickness under ultrasound in people with AIS, did not see a difference in transverse abdominus muscle activation between individuals with scoliosis and a healthy control group during rest, but they reported a significant difference between both groups during contraction. Although abdominal muscle thickness has been evaluated in individuals with scoliosis in the literature, there is no study in the literature reporting the relationship between abdominal muscle thickness under ultrasound as a result of schroth exercises. The aim of this study is to evaluate the effectiveness of the Schroth method on abdominal muscle thickness in people with AIS.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with idiopathic scoliosis by a specialist physician,
* 10-18 years old,
* The primary curvature is between 10-45 degrees according to the Cobb method,
* C or S scoliosis,
* Pain in the back/lumbar region due to scoliosis,
* Those who have not received any exercise therapy for scoliosis before,
* Volunteer to participate in the study,
* Having the cognitive capacity to cooperate with the guidance of the physiotherapist,
* Have not had any musculoskeletal injury in the last 6 months,
* No neurological, orthopedic or cardiopulmonary disorders other than the diagnosis of scoliosis,
* Young individuals who have not undergone any surgery related to the diagnosis of scoliosis will be included in the study.

Exclusion Criteria:

* The patient has any contraindications for exercise,
* Having had previous spine surgery and abdominal surgery,
* Having any mental problems,
* The fact that scoliosis is not idiopathic but has arisen for different reasons (neurological, congenital),
* In case of neurological, psychiatric, muscular, rheumatic or orthopedic diseases, these people will not be included in the study.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2023-06-08 (Estimated); Study Completion 2023-09-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of Abdominal Muscle Thickness Measurement Under Ultrasound | 6 weeks
  Abdominal muscle imaging and measurement will be performed with the participants lying on their back with the soles of the feet on the bed with the knees flexed to 90 degrees and the hips to approximately 45 degrees of flexion. The medial convex probe will be placed at the intersection point of a horizontal line drawn from the navel to the lateral and a vertical line drawn from the anterior superior iliac spine to the cranial. The probe will be placed transversely so that the medial fascia of the transversus abdominus is medial to the image and the transversus abdominus, internal oblique and external oblique muscles are well visible.

SECONDARY OUTCOMES:
Assessment of Risser Sign | 6 weeks
  The epiphyseal plate starts from the lateral border of the anterior superior spina iliaca, moves medially, and ends at the posterior superior spina iliaca. The degree of completion is expressed as a percentage: Grade 1 ≤ 25%, Grade 2 26-50%, Grade 3 51-75%, Grade 4 75-100%. When the epiphysis is combined with the illium, it is defined as Grade 5. The Risser sign is used to determine the age of bone development, growth rate and risk level for scoliosis. In the study, it was used to determine the age of bone development. It has been reported to be reliable and sensitive in determining the age of bone development.
Assessment of cobb angle | 6 weeks
  The degree of curvature in the coronal plane is measured radiographically according to the Cobb method. The Cobb angle, considered the gold standard, is the angle between the perpendiculars when descending lines drawn from the top of the curve along the upper endplate of the most tilting vertebra at the top and the lines drawn under the lower endplate of the most tilting vertebrae to the bottom. The Cobb angle describes only one plane of a three-dimensional deformity, but provides information about the progression of the curvature. Observer variability was recorded as 2.8°-4.9° and interobserver variability was recorded as 6.3°-7.2° in Cobb angle measurement with conventional techniques. In digital Cobb angle measurements, the variability for the same observer and the interobserver variability were reported as 1.3°. In the study, it is planned to evaluate the Cobb angle by the relevant physician.
Assessment of Angle of Trunk Rotation | 6 weeks
  Measurement of trunk rotation angle/degree is the most appropriate method used in the clinical evaluation of scoliosis. ATR can be used to monitor the effects of treatment without radiographic evaluation. ATR measurement is done using a special inclinometer called a scoliometer. The patient is asked to lean forward with the arms relaxed. The scoliometer is placed posteriorly and the degree observed at the point of greatest gibbosis is recorded. ATR is a reliable measurement with a repeatability of 86%. A variation of 2° in interobserver measurements can be considered significant. In this study, it is planned to evaluate ATR measurements before and after treatment with a Scoliometer® brand scoliometer. There is a correlation between the Scoliometer® and the Cobb angle. The Scoliometer® has been observed to have specificity, sensitivity and predictive ability. Intra-rater and inter-rater reliability coefficients are r = .86-.97
Assessment of Quality of Life | 6 weeks
  Disease-related quality of life of young individuals included in the study, Alanay A. et al. It will be evaluated with the Scoliosis Research Society 22. Form (SRS 22r) scale, developed by the Scoliosis Research Society, which has been translated into Turkish and has proven validity and reliability. Scale "Which of the following answers best describes the pain you have experienced during the past 6 months?", "How much are you able to move now?", "How long have you felt calm and peaceful during the last 6 months?" It consists of 22 questions and 5 sub-dimensions. Sub dimensions; pain, self-image/view, spinal functions, mental health, and satisfaction with treatment. All of these sections are evaluated separately and/or all questions are collected under the total score. High scores indicate high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Zeynep Ayyıldız Eroğlu, Istanbul, Bahcelievler, Turkey (Türkiye)

REFERENCES:
- [Background] Schreiber S, Parent EC, Khodayari Moez E, Hedden DM, Hill DL, Moreau M, Lou E, Watkins EM, Southon SC. Schroth Physiotherapeutic Scoliosis-Specific Exercises Added to the Standard of Care Lead to Better Cobb Angle Outcomes in Adolescents with Idiopathic Scoliosis - an Assessor and Statistician Blinded Randomized Controlled Trial. PLoS One. 2016 Dec 29;11(12):e0168746. doi: 10.1371/journal.pone.0168746. eCollection 2016. PMID 28033399
- [Background] Rigo M, Reiter Ch, Weiss HR. Effect of conservative management on the prevalence of surgery in patients with adolescent idiopathic scoliosis. Pediatr Rehabil. 2003 Jul-Dec;6(3-4):209-14. doi: 10.1080/13638490310001642054. PMID 14713587